CLINICAL TRIAL: NCT06678854
Title: First Responder Aphasia Strategy Training
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2024-1447; A481800 (Other: UW Madison); Protocol Version Oct 2024 (Other: UW Madison)
Record Dates: First submitted 2024-11-04; First posted 2024-11-07 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Aphasia
MeSH Terms: conditions — Aphasia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- First Responders (Experimental)
  Interventions: Other: Training about Aphasia

INTERVENTIONS:
Other: Training about Aphasia — Training will include direct teaching, aphasia simulations, scenario-based training and a panel with persons with aphasia with the goal of increasing confidence for law enforcement officers and first responders providing services to and communicating with persons with aphasia.

SUMMARY:
This study aims to determine the impact of a collaborative approach to training law enforcement officers and first responders about aphasia including their knowledge and confidence in communicating with individuals with aphasia that they may encounter in the field. 75 participants from Madison Police Department will be enrolled and can expect to be on study for up to 6 months.

DETAILED DESCRIPTION:
The investigators will partner with the Madison Police Department to provide training and programming to law enforcement officers and first responders. Training will include direct teaching, aphasia simulations, scenario-based training and a panel with persons with aphasia with the goal of increasing confidence for law enforcement officers and first responders providing services to and communicating with persons with aphasia.

Participants will take 3 surveys over 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Employed by Madison Police Department as a first responder or law enforcement officer
* willing and able to provide informed consent
* willing to comply with all study procedures and be available for the duration of the study

Exclusion Criteria:

* Not employed as a first responder or law enforcement officer with Madison Police Department

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2024-11-05 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
First Responder Aphasia Training Score | pre-test (baseline), post-test (after 1 day of training)
  Two items scored from 1 (very confident) to 4 (not confident) where lower scores indicate increased confidence in communication with a person with Aphasia.
First Responder Aphasia Training Score | pre-test (baseline), 3 to 6 month follow-up
  Two items scored from 1 (never), 2 (a few times), 3 (regularly), 4 (I'm not sure) about whether they have interacted with a person with Aphasia in their professional and personal lives.
First Responder Strategies for Aphasia | pre-test (baseline), post-test (after 1 day of training), 3 to 6 month follow-up
  First responders are to list 10 strategies for competence, understanding, and expression in communicating with a person with Aphasia. Count of correct strategies will be reported.
First Responder Confidence in Communication Score | pre-test (baseline), post-test (after 1 day of training), 3 to 6 month follow-up
  Scored from 1 (very uncomfortable) to 5 (very comfortable), with higher scores indicating higher confidence.

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Mueller, PhD, CCC-SLP, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No